CLINICAL TRIAL: NCT04828200
Title: Multi-Dimensional Evaluation Of The Presence Of Sarcopenia In Patients With Knee Osteoarthritis
Brief Title: The Presence Of Sarcopenia In Patients With Knee Osteoarthritis
Status: Completed | Type: Observational
Sponsor: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Sefa Gümrük Aslan, Physical Medicine and Rehabilitation Specialist, Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Other Study IDs: 2
Record Dates: First submitted 2021-03-28; First posted 2021-04-01 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Sarcopenia; Osteoarthritis
Keywords: Dual-X-ray absorptiometry; Sarcopenia; Knee osteoarthritis; ultrasonography
MeSH Terms: conditions — Sarcopenia; Osteoarthritis; Osteoarthritis, Knee | interventions — Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- sarcopenic patints with knee ostheoarthritis: 12 patients between the ages of 50-70, who have been followed up with the diagnosis of knee Ostheoarthritis (OA) patients with sarcopenia.All subjects were evaluated by the European Working Group on Sarcopenia in Older People (EWGSOP) diagnostic criteria for the diagnosis of sarcopenia.
  Interventions: Diagnostic Test: Musculoskeletal ultrasound; Diagnostic Test: Dual-X-ray absorptiometry; Diagnostic Test: Isokinetic dynamometer
- non sarcopenic patients with knee ostheoarthritis: 90 patients between the ages of 50-70, who have been followed up with the diagnosis of knee Ostheoarthritis (OA) patients.
  Interventions: Diagnostic Test: Musculoskeletal ultrasound; Diagnostic Test: Dual-X-ray absorptiometry; Diagnostic Test: Isokinetic dynamometer
- control group: 33 patients between the ages of 50-70, who have been followed up not being exposed to be sarcopenia or knee OA
  Interventions: Diagnostic Test: Musculoskeletal ultrasound; Diagnostic Test: Dual-X-ray absorptiometry; Diagnostic Test: Isokinetic dynamometer

INTERVENTIONS:
Diagnostic Test: Musculoskeletal ultrasound — The ultrasonographic assesment will be used to examine the rectus femoris, gastrocnemius medailalis and rectus abdominis subcutaneous and muscle thickness. Additionally, fascicle length and pennation angle were measured between the two parallel aponeuroses of the gastrocnemius muscle (bulkiest part of medial head) in the longitudinal view when subjects were in prone position with their ankles at 90°.
Diagnostic Test: Dual-X-ray absorptiometry — The muscle masses of the patients were evaluated by measuring the fat mass (Fat Mass-FM), fat mass index (FMI), lean body mass (LBM) and skeletal muscle index (SMI) calculated by DEXA. Appendicular muscle mass (ASM) is calculated by summing the lean soft tissue of the two upper limbs and the two lower limbs. Skeletal muscle mass index is calculated by dividing the appendicular lean mass by the square of the neck height [SMI = ASM / height2 (kg / m2)].
Diagnostic Test: Isokinetic dynamometer — Quadriceps-hamstring Peak Torque (PT) values and the ratio of PT values to body weight (PT / VA) (at 60 and 180 ° / sec speeds) were evaluated with an isokinetic dynamometer

SUMMARY:
Osteoarthritis (OA) is one of the most common joint disorders worldwide . The knee is the most common symptomatic joint in osteoarthritis. In this study, we evaluated the presence of sarcopenia multidimensionally in patients with knee osteoarthritis (OA) using clinical, ultrasonographic and biochemical parameters, and in this respect, it was aimed to investigate the relation between OA and sarcopenia and to identify the most practical, easily accessible and inexpensive method for investigating sarcopenia.

DETAILED DESCRIPTION:
102 patients with clinical and radiological diagnosis of knee osteoarthritis and 33 healthy control subjects were included in the study. A total of 135 subjects were evaluated using the European Working Group on Sarcopenia in Older People (EWGSOP) diagnostic criteria of sarcopenia. The first group consists of (OA) patients with sarcopenia, the second group consist of OA patients without sarcopenia and the third group is controls subjects. The detailed musculoskeletal system examination of the patients included in the study was carried out by a single physician, and complete blood count, renal function tests, electrolytes, total protein, albumin, 25 (OH) vitamin D, serum leptin, serum adiponectin, PTH, TSH and vitamin B12 values were recorded using the venous blood samples taken from the study group.Dual-X-ray absorptiometry (DEXA) is used to measure Body composition parameters and muscle mass measurements, isometric muscle strength evaluations, handgrip strength and gait speeds for diagnosis of sarcopenia. Short-form -36 (SF-36) The Nutritional Assessment-short form (MNA), the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), the International Physical Assessment Questionnaire Short Form (IPAQ-SF) and the Center for Epidemiologic Studies Depression Scale (CES-D scale) were administered to every patient as outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 50-70

  * Patients who have been followed up with the diagnosis of knee ostheoarthritis
  * Patients who have been followed up with the diagnosis of knee ostheoarthritis and sarcopenia

Exclusion Criteria:

* Previous history of any trauma/surgical history of the lower extremities (other than amputation)
* Rheumatic diseases Contracture of the knee and the ankle of the intact limb
* malignant disease
* hyperthyroidism/ hypothyroidism
* chronic inflammatory disease
* diabetes mellitus, and uncontrollable heart and kidney diseases
* pregnant women

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 102 patients ages 50 to 70 years were diagnosed with knee osteoarthritis according to the American College of Rheumatology criteria and 33 healthy volunteers were enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2016-04-10 (Actual); Primary Completion 2016-09-10 (Actual); Study Completion 2016-09-10 (Actual)

PRIMARY OUTCOMES:
Musculoskeletal ultrasonography | through study completion, an average of one and a half months
  Rectus femoris, Rectus abdominis and gastrocnemius subcutaneosus and muscle thickness measurements will be performed by using ultrasound.

SECONDARY OUTCOMES:
The Western Ontario and McMaster Universities Arthritis Index (WOMAC) | through study completion, an average of one and a half months
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) is a widely used, proprietary set of standardized questionnaires used by health professionals to evaluate the condition of patients with osteoarthritis of the knee and hip, including pain, stiffness, and physical functioning of the joints. The test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4).
  The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. The WOMAC is scored on a best to worst scale, so that lower subscale scores represent less pain, less stiffness, or better physical function.
Short Form-36 (SF-36) | through study completion, an average of one and a half months
  The health-related quality of life of the subjects will be evaluated with Short Form-36 (SF-36). This comprises 36 questions related to eight different subscales, physical functioning, bodily pain, role limitation, due to physical health problems, general health perceptions, vitality, energy and fatigue, role limitations due to emotional problems, social functioning and general mental health, which covers psychological distress and wellbeing. Each of eight subscales is scored between 0 and 100, with higher scores indicating a better quality of life.
The Center for Epidemiologic Studies Depression Scale (CES-D scale) | through study completion, an average of one and a half months
  The CES-D scale is a brief self-report scale designed to measure self-reported symptoms associated with depression experienced in the past week. The items of the scale are symptoms associated with depression which have been used in previously validated longer scales. TheCES-D contains 20 items that can be responded to on a four-point Likert scale, with response categories ranging from 'rarely or none of the time' (0 points) to 'most or all of the times' (3 points) which are summed up to a total score where higher score indicate more severe depressive symptoms. A cut-off score of ≥ 16 is generally accepted as indicator for clinical meaningful depressive symptoms.
The timed 'Up & Go' test | through study completion, an average of one and a half months
  The Timed Up and Go test (TUG) is a simple test used to assess a person's mobility and requires both static and dynamic balance. It uses the time that a person takes to rise from a chair, walk three meters, turn around 180 degrees, walk back to the chair, and sit down while turning 180 degrees.
International Assessment Questionnaire Short Form (IPAQ-SF) | through study completion, an average of one and a half months
  This measure assesses the types of intensity of physical activity and sitting time that people do as part of their daily lives are considered to estimate total physical activity in MET-min/week and time spent sitting. 2 METS is twice what you expend at rest. Data collected with IPAQ can be reported as a continuous measure and reported as median METminutes. Median values can be computed for walking (W), moderate-intensity activities (M), and vigorous-intensity activities (V) using the following formulas: Walking MET-minutes/week = 3.3 * walking minutes * walking/days, Moderate MET-minutes/week = 4.0 * moderate-intensity activity minutes * moderate days Vigorous MET-minutes/week = 8.0 * vigorous-intensity activity minutes * vigorous-intensity days.
Mini-Nutritional Assessment (MNA-SF) | through study completion, an average of one and a half months
  The MNA® is a validated nutrition screening and assessment tool that can identify geriatric patients age 65 and above who are malnourished or at risk of malnutrition.

CONTACTS AND LOCATIONS:
Overall Officials: Sefa gümrük aslan, Principal Investigator — Gaziler Physical Medicine And Rehabilitation Health Application And Research Center
Locations (1):
- Gaziler PMR, Training and Research Hospital, Department of PMR, Ankara, Çankaya/turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No